CLINICAL TRIAL: NCT02642601
Title: Role of Indomethacin in Cases of Difficult Embryo Transfer in Intra Cytoplasmic Sperm Injection Cycles
Brief Title: Role of Indomethacin in Difficult Embryo Transfer.
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mona M Shaban, Dr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MS62014
Record Dates: First submitted 2015-12-24; First posted 2015-12-30 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Difficult Embryo Transfer
Keywords: indomethacin, ICSI, difficult embryo transfer
MeSH Terms: interventions — Indomethacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- indomethacin (Experimental): one dose of indomethacin 100 mg rectal suppository;will be adminstrated1-2 hours before embryo transfer
  Interventions: Drug: Indomethacin(KAHIRA PHARMA&CHEM,IND,CO.CAIRO-EGYPT)
- no medication (No Intervention): no indomethacine before embryo transfer

INTERVENTIONS:
Drug: Indomethacin(KAHIRA PHARMA&CHEM,IND,CO.CAIRO-EGYPT) — one dose of indomethacin 100 mg rectal suppository 1- 2 hours before embryo transfer
  Other Names: indocid
  Arms: indomethacin

SUMMARY:
the aim of the study is to assess the role of indomethacin in cases of difficult embryo transfer in intracytoplasmic sperm injection cycles.

DETAILED DESCRIPTION:
It is a prospective randomized study in which 200 women undergoing ICSI( intracytoplasmic sperm injection) and fulfilling the inclusion criteria(Difficult mock embryo transfer on day of ovum pick up ,Women's age 20-38 yaears,Early follicular FSH ≤10 IU/l ,Tubal, male infertility, unexplained factors of infertility.) will be recruited.

All patients will received long stimulation protocol ;down regulation will be achieved by administration of triptorelin0.1 mg(decapeptyl 0.1 mg, Ferring, Malmo, sweden) S.C daily from day 21 of the cycle preceding the stimulation cycle till the day of hCG administration.,down regulation will be checked day 2 of stimulation cycle by checking serum E2˂50 pg/ml, endometrial thickness ˂ 5mm and quiescent both ovaries.

When down regulation is achieved stimulation is commenced using hmG(Menogon, ferring pharmaceuticals, Germany) 225 IU daily intramuscular injection, Serial trans-vaginal ultrasound to assess follicular growth and serum E2 are done starting on day 6 of the cycle and onward, with adjustments of gonadotropin dose and monitoring frequency based on patient response.

Once 3 or more leading follicles reached≥18mm hCG 10000 IU (Pregnyl; NV Organon) will be administrated IM.

Ovum pick up will be done 34-36 hours following hCG administration with ultrasound guidance under general anesthesia.after that mock embryo transfer will be done using labotec embryo transfer catheter and women in which any degree of difficulty according to Tomas et al. 2002 criteria will be recruited in the study and divided randomly into two groups according to computer generated random cards ;group A (n=100): will receive indomethacin 100 mg rectal supp(KAHIRA PHARMA&CHEM,IND,CO.CAIRO-EGYPT) 1-2 hours before embryo transfer, group B (n=100) will not receive any medications before embryo transfer.

Embryo transfer of 2 embryos will be done by the same technique in lithotomy position with full bladder under ultrasound guidance 2-3 days after ovum pick up depending on the number and quality of available embryos using labotec catheter (Labotec, Gottingen Germanny).

Luteal phase will be achieved Using progesterone vaginal pessaries (Cyclogest, Alpharma, UK) 400 mg twice daily from the day of egg collection till the day of the pregnancy test and continued till 12 week gestation if pregnancy is documented.

ELIGIBILITY:
Inclusion Criteria:

* Infertile patients undergoing ICSI cycle with difficult mock transfer done on day of day of ovum pick up

Exclusion Criteria:

* repeated ICSI failure
* Easy mock embryo transfer on day of ovum pick up
* Early follicular FSH >10 IU/l
* Past history of allergy to NSAID.
* Past history of asthma, peptic ulcer disease or inflammatory bowel disease. Endometrial pathology

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-12 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy rate | 2 weeks after +ve pregnancy test
  +ve pregnancy test+ gestational sac with fetal pulsation by ultrasound

SECONDARY OUTCOMES:
Implantation rate | the number of total gestational sacs divided by the total number of embryos transferred.
  2-4 weeks after positive pregnancy test

OTHER OUTCOMES:
ongoing pregnancy rate | after 12 weeks gestation
  pregnancy exceeding 12 weeks gestation

CONTACTS AND LOCATIONS:
Overall Officials: Mona M Shaban, MD, Principal Investigator — Cairo University
Locations (2):
- Egypt (2):
  - IVF center,Cairo university hospital,Egypt, Cairo
  - Kamal Shoeir private IVF center,Cairo,Egypt, Cairo